CLINICAL TRIAL: NCT01439646
Title: Observational, Retrospective Study to Evaluate the Clinical Outcome in High Risk Patients Who Received Empirical Antifungal Therapy
Brief Title: Study to Evaluate the Clinical Outcome in High Risk Patients Who Received Empirical Antifungal Therapy
Status: Completed | Type: Observational
Sponsor: Fortis Hospital, India (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr Raja Dhar, Consultant Pulmonologist, Fortis Hospital, India
Other Study IDs: Rdhar India
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Antifungal Therapy
Keywords: empirical; ICU; high risk patient

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non neutropenic, ICU, empiric ,antifungals
  Interventions: Other: it is a retrospective study, hence no active intervention

INTERVENTIONS:
Other: it is a retrospective study, hence no active intervention — since it is an observational restrospective study hence no active intervention is planned

SUMMARY:
Retrospective, observational study To study the effect of Empirical Antifungal therapy on clinical outcome in high risk patients with suspected Invasive Fungal Infection admitted in ICU/Critical care unit, To know the current epidemiology of IFI and management approach in patients at high risk of Invasive fungal infections, Identify the risk factors associated with Invasive fungal infections, To comment on the appropriateness of empirical therapy used based on proven/probable diagnosis

DETAILED DESCRIPTION:
Study Objectives

Primary Objective:

- To study the effect of Empirical Antifungal therapy on clinical outcome in high risk patients with suspected Invasive Fungal Infection admitted in ICU/Critical care unit

* Secondary Objectives:

  1. To know the current epidemiology of IFI and management approach in patients at high risk of Invasive fungal infections
  2. Identify the risk factors associated with Invasive fungal infections
  3. To comment on the appropriateness of empirical therapy used based on proven/probable diagnosis

     Inclusion criteria:

     All Non-neutropenic patients admitted in the intensive care/critical care unit who are prescribed any form of pre-emptive / empirical Antifungal therapy during the specified study duration period

     Exclusion criteria:

     Neutropenic patients Patients with proven invasive fungal infections where antifungal therapy was initiated after the confirmation of Invasive fungal infection/Candidemia Patients who received prophylactic antifungal agents

     Study Design
* Multi Center (Dual-center - Fortis Hospital and Apollo Hospital) Retrospective, Observational Study
* Study Patients: 100 in number

Retrospective data will be collected for all patients admitted in intensive care unit/Critical care unit (under the study investigators) who received any form of Empirical / Preemptive (not prophylactic) Antifungal therapy (of any duration, irrespective of culture positivity) as a suspected case of Invasive Fungal Infection.

Following details of patients will be captured

Demographics, primary and secondary diagnosis, co-morbidities, grade of infection, severity of sepsis and disease.

Daily hemodynamic parameters, routine blood tests including Total count and hematologic profile, renal profile, Liver function tests, electrolyte status, additional tests whatever was done as a course of the therapy.

Fungal C/S reports and any other sample culture reports

Duration of treatment, Changes in therapy, Adjuvant therapy - for relevant cases, Any Surgical procedures undertaken: e.g., surgical debridement, fasciotomy and dressing (as a part of the standard treatment according to available guidelines) - for relevant cases, Any additional invasive procedure (eg: Mechanical ventilation ), Reported adverse events

Recording of Risk factors for invasive fungal infections as detailed but not limited to:

1. Diabetes,
2. Use of immunosuppressants (Eg. steroids)
3. Chronic Hemodialysis , TPN, Mechanical ventilation ,
4. Sepsis/Septic shock, Multiorgan dysfunction (more than one organ),
5. Non response to > 4 days of broad spectrum antibiotics,
6. Structural lung disease,
7. Major abdominal surgery,
8. Multifocal colonization

   * Study Duration:

A period of one year starting backwards from December 2010 till January 2010.( max. 100 patients retrospectively tracking back from Dec 2010 whichever comes first ).

Statistical analysis

Appropriate statistical tools such as "Multiple logistic regressions" model will be used to analyze linkages between different parameters recorded in the study

Primary Endpoint:

1. Mortality both Short term (while on antifungal therapy) and Long term (within 12 weeks of completion of antifungal therapy)
2. Mean Duration of ICU (Intensive Care Unit) / HDU (High Dependency Unit stay after initiation of Antifungal Therapy

Secondary Endpoints:

The common pathogens associated with Invasive Fungal Infections

The common empirical antifungal agents used in suspected Invasive Fungal Infection

The mean time for initiation of Antifungal therapy after suspicion of invasive fungal infection.

The mean duration of antifungal therapy

The risk factors in patients with proven/probable invasive fungal infections

The appropriateness of antifungal agent based on microbiological and/or clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* All Non-neutropenic patients (18-75yrs) admitted in the intensive care/critical care unit who are prescribed any form of pre-emptive / empirical Antifungal therapy during the specified study duration period

Exclusion Criteria:

* Neutropenic patients
* Patients with proven invasive fungal infections where antifungal therapy was initiated after the confirmation of Invasive fungal infection/Candidemia
* Patients who received prophylactic antifungal agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients , nonneutropenic in ICU who have risk factors for fungal infections and are started empiricaly on antifungals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Mortality both Short term (while on antifungal therapy) and Long term (within 12 weeks of completion of antifungal therapy) | 6 months
Mean Duration of ICU (Intensive Care Unit) / HDU (High Dependency Unit stay after initiation of Antifungal Therapy | 6 months

SECONDARY OUTCOMES:
The common pathogens associated with Invasive Fungal Infections | 6 months
The common empirical antifungal agents used in suspected Invasive Fungal Infection | 6 months
The mean time for initiation of Antifungal therapy after suspicion of invasive fungal infection | 6 months
The risk factors in patients with proven/probable invasive fungal infections | 6 months
The appropriateness of antifungal agent based on microbiological and/or clinical outcome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: raja dhar, MD, Principal Investigator — Fortis Hospital, Kolkata
Locations (1):
- Raja dhar, Kolkata, West Bengal, India